CLINICAL TRIAL: NCT05763914
Title: Hand Eczema in Cleaners: a Randomized Clinical Trial of Picture-based Prevention Compared to Treatment as Usual Among Professional Hospital Cleaners
Brief Title: A 24-week Single-blind Trial of Prevention of Hand Eczema in Cleaners
Acronym: HEIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: University of Copenhagen (Other); Danish Working Environment Fund (Unknown)
Responsible Party: Principal Investigator, Farnam Barati Sedeh, Principal Investigator, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20205100702
Record Dates: First submitted 2023-02-14; First posted 2023-03-10 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Hand Eczema
Keywords: Prevention; Occupational; Picture; Cleaning

STUDY DESIGN:
Intervention Model Description: A cluster-randomized clinical trial, including three different hospitals. At each hospital, 78 cleaners will be included.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Picture-based prevention education and an educational course (Experimental): The participants will have access to picture-based prevention education, and at the same time, they will participate in an educational course.
  Interventions: Behavioral: Change in the incidence of hand eczema; Behavioral: Change in severity of hand eczema; Behavioral: Change in the number of self-reported days with absence from work due to having hand eczema; Behavioral: Change in the number of participants being forced to change their job due to having hand eczema; Behavioral: Change in The Quality Of Life in in relation to hand eczema; Behavioral: Change in the level of knowledge regarding skin care and protection.
- Group 2: Picture-based prevention education only (no educational course) (Experimental): The participants will only have access to picture-based prevention education and will not participate in any educational course.
  Interventions: Behavioral: Change in the incidence of hand eczema; Behavioral: Change in severity of hand eczema; Behavioral: Change in the number of self-reported days with absence from work due to having hand eczema; Behavioral: Change in the number of participants being forced to change their job due to having hand eczema; Behavioral: Change in The Quality Of Life in in relation to hand eczema; Behavioral: Change in the level of knowledge regarding skin care and protection.
- Group 3: Placebo (control) (Placebo Comparator): The participants will not have access to picture-based prevention education and do not participate in any educational course.
  Interventions: Behavioral: Change in the incidence of hand eczema; Behavioral: Change in severity of hand eczema; Behavioral: Change in the number of self-reported days with absence from work due to having hand eczema; Behavioral: Change in the number of participants being forced to change their job due to having hand eczema; Behavioral: Change in The Quality Of Life in in relation to hand eczema; Behavioral: Change in the level of knowledge regarding skin care and protection.

INTERVENTIONS:
Behavioral: Change in the incidence of hand eczema — Assessed by the self-reported cases of newly-developed hand eczema. Change between baseline and 6 months.
Behavioral: Change in severity of hand eczema — Assessed by using the Hand Eczema Severity Index (HECSI). HECSI score: 0-360 points (0 best, 360 worst). Change between baseline and 6 months.
Behavioral: Change in the number of self-reported days with absence from work due to having hand eczema — Self-reported total number of sick days due to having hand eczema. Change between baseline and 6 months.
Behavioral: Change in the number of participants being forced to change their job due to having hand eczema — Self-reported change of job due to having hand eczema. Change between baseline and 6 months.
Behavioral: Change in The Quality Of Life in in relation to hand eczema — Assessed by using Hand Eczema Questionnaire (QolHEQ). Change between baseline and 6 months.
Behavioral: Change in the level of knowledge regarding skin care and protection. — Self-reported level of knowledge regarding skin care and protection. Change between baseline and 6 months.

SUMMARY:
This study aims to investigate the effectiveness of picture-based prevention education among professional hospital cleaners in relation to hand eczema. This is a single-blinded randomized clinical trial including hospital cleaners at three different hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Professional hospital cleaners ≥ 18 years old
* Sufficient Danish skills
* Written informed consent

Exclusion Criteria:

* Insufficient Danish skills
* Pregnancy
* Other skin diseases on the hands
* Receiving Immunomodulatory therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-06-24 (Actual); Study Completion 2023-06-24 (Actual)

PRIMARY OUTCOMES:
Incidence rate of hand eczema | Change between baseline and 6 months
  Measured by a self-reported questionnaire
Hand Eczema Severity Index (HECSI) | Change between baseline and 6 months
  Objective assessment of disease severity, measured by HECSI-score: 0-360 points (0 best, 360) worst)

SECONDARY OUTCOMES:
Rate of absence from work due to having hand eczema | Change between baseline and 6 months
  Measured by a self-reported questionnaire
Rate of participants being forced to change their job due to having hand eczema (questionnaire-based). | Change between baseline and 6 months
  Measured by a self-reported questionnaire
The Quality Of Life in Hand Eczema Questionnaire (QqlHEQ) | Change between baseline and 6 months
  Subjective assessment of quality of life using QqlHEQ which contains 30 items; generally, all items are scored 0-4 (only three items differ in their scoring structure).
Rate of knowledge regarding skin care and protection. | Change between baseline and 6 months
  Measured by a self-reported questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Sophie Ibler, M.D., Principal Investigator — Zealand University Hospital
Locations (1):
- Cleaning departments at Køge, Slagelse and Holbæk hospitals, Køge, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The results of the project will be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Materials will be made available six months after the publication of the primary outcomes.